CLINICAL TRIAL: NCT02778503
Title: Effectiveness of Atraumatic Restorative Treatment Using Glass Ionomer Cement of Different Costs: a Randomized Controlled Trial
Brief Title: Effectiveness of Atraumatic Restorative Treatment Using Glass Ionomer Cement of Different Costs
Acronym: SLM1797
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty Sao Leopoldo Mandic Campinas (Other)
Responsible Party: Principal Investigator, Jose Carlos P Imparato, PhD, Senior Lecturer, Faculty Sao Leopoldo Mandic Campinas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SLM2
Record Dates: First submitted 2016-04-07; First posted 2016-05-20 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Dental Caries
Keywords: Tooth, Deciduous; Dentition, Permanent; Dental Atraumatic Restorative Treatment; Glass Ionomer Cements; Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Technology, High-Cost

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Cost (Active Comparator): Restoration using a high-cost glass ionomer cement.
  Interventions: Other: High Cost
- Low Cost (Experimental): Restoration using a low-cost glass ionomer cement.
  Interventions: Other: Low Cost

INTERVENTIONS:
Other: High Cost — Surfaces allocated to this group will be treated with a high-cost glass ionomer cement restoration (Fuji IX, GC America, USA), according to the manufacturer's instructions.
  Arms: High Cost
Other: Low Cost — Surfaces allocated to this group will be treated with a low-cost glass ionomer cement restoration (Maxxion R, FGM, BRA), according to the manufacturer's instructions.
  Arms: Low Cost

SUMMARY:
Atraumatic Restorative Treatment (ART) is an alternative restorative technique for dental caries, applying the partial caries tissue removal philosophy using hand instruments, relative cotton rolls isolation, immediate restoration with Glass Ionomer Cements (GIC) and avoiding local anesthesia. The chosen material for this study will be the High Viscosity Glass Ionomer Cement (HVGIC) due to its unique physical-chemical properties as well as its applicability in challenging clinical situations where other materials would not be adequate. Although there are substantial evidences regarding GIC properties, information about GIC (with different costs) longevity is still weak. Therefore, the objective of this study is to assess the effectiveness of ART restorations performed with low-cost HVGIC in cavitated dentine carious lesions in primary and permanent molars. This will be a multicenter randomized controlled double-blind (patient and operator) clinical trial performed with 680 primary and/or permanent molars in children between 4 and 9 years old presenting cavitated dentine carious lesions in occlusal and occlusal-proximal surfaces. The tooth will be considered as the unit sample, which will be randomly allocated to the groups through a generated random list numbers and distributed in dark sealed envelopes opened only by dental assistants. Teeth in the test group will be submitted to restorative treatment with HVGIC Vitro Molar and those in the control group with HVGIC Fuji IX. The restoration effectiveness will be assessed by means of both clinical and bitewing x-rays control after 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Children with at least one primary and/or permanent molar with dentine carious lesion in the occlusal and/or occlusal-proximal surface.

Exclusion Criteria:

* Special need patients, subjects under orthodontic treatment and/or systemically compromised.
* Teeth with restorations, sealants, developmental defects, deep carious lesions with pulpal exposure risk, fistula and/or abscess, and those with history of spontaneous pain.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 574 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Restoration survival | 12 months
  The restoration will be classified according to the scores described by Frencken et al. (1994) and Roeleveld et al. (2006).

SECONDARY OUTCOMES:
Cost-effectiveness | Through study completion (12 months)
  The costs of each treatment procedure will be calculated and compared with thresholds values for intervention cost-effectiveness by region, determined by World Health Organization (http://www.who.int/choice/costs/CER_levels/en/).
Impact on children's quality of life | Baseline and 12 months
  The oral health related quality of life will be measured using a validated questionnaire according to the children's age. The "Early Childhood Oral Health Impact Scale" (ECOHIS) (Tesch et al., 2008) will be applied with 4-5 years old children. The "Child Perceptions Questionnaire" (CPQ) will be used for 6-9 years old children (Martins et al., 2009). They will be applied immediately before the procedure and on 12 months follow-up.
Children self-reported discomfort | Baseline
  The discomfort of each treatment will be evaluated using the facial scale of Wong-Baker (Wong, Baker, 1988). The patient will be asked to choose the face that is more similar to how he/she felt during the treatment. The answer should be given solely by the child, which means no parental or professional interferences.
Caries lesions progression | Every 6 months up to 12 months
  The treatments will be evaluated radiographically. This evaluation will be performed by two blinded examiners, which will evaluate the four patients' radiographies (baseline, after treatment, 6 months, 12 months) independently, two by two, without knowing the chronological order of them. The efficacy of the treatment will be related to the presence or absence of increasing radiolucent area. They will also classify each radiography using Ekstrand criteria (Ekstrand et al., 1997) and analyze them in a software (ImageJ 1.49, National Institute of Health, USA) in order to make the radiographic subtraction.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Carlos P Imparato, PhD, Principal Investigator — Faculty Sao Leopoldo Mandic
Locations (1):
- Faculty Sao Leopoldo Mandic, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ekstrand KR, Ricketts DN, Kidd EA. Reproducibility and accuracy of three methods for assessment of demineralization depth of the occlusal surface: an in vitro examination. Caries Res. 1997;31(3):224-31. doi: 10.1159/000262404. PMID 9165195
- [Background] Frencken JE, Pilot T, Songpaisan Y, Phantumvanit P. Atraumatic restorative treatment (ART): rationale, technique, and development. J Public Health Dent. 1996;56(3 Spec No):135-40; discussion 161-3. doi: 10.1111/j.1752-7325.1996.tb02423.x. PMID 8915958
- [Background] Martins MT, Ferreira FM, Oliveira AC, Paiva SM, Vale MP, Allison PJ, Pordeus IA. Preliminary validation of the Brazilian version of the Child Perceptions Questionnaire 8-10. Eur J Paediatr Dent. 2009 Sep;10(3):135-40. PMID 19761288
- [Background] Roeleveld AC, van Amerongen WE, Mandari GJ. Influence of residual caries and cervical gaps on the survival rate of Class II glass ionomer restorations. Eur Arch Paediatr Dent. 2006 Jun;7(2):85-91. doi: 10.1007/BF03320820. PMID 17140533
- [Background] Tesch FC, Oliveira BH, Leao A. [Semantic equivalence of the Brazilian version of the Early Childhood Oral Health Impact Scale]. Cad Saude Publica. 2008 Aug;24(8):1897-909. doi: 10.1590/s0102-311x2008000800018. Portuguese. PMID 18709230
- [Background] Wong DL, Baker CM. Pain in children: comparison of assessment scales. Pediatr Nurs. 1988 Jan-Feb;14(1):9-17. No abstract available. PMID 3344163